CLINICAL TRIAL: NCT05409677
Title: Perioperative Eosinophils And Their Recovery Serve As Prominent Predictors For Type A Acute Aortic Dissection Prognosis
Brief Title: Perioperative Eosinophils Their Recovery in Type A Acute Aortic Dissection Prognosis
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: 81871607
Record Dates: First submitted 2022-05-25; First posted 2022-06-08 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-05

CONDITIONS: Acute Aortic Dissection
Keywords: Type A acute aortic dissection; Eosinophils; Prognosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1-month survivors; 1-month non-survivors: Depending on mortality within 1 month, the patients were divided into two groups named 1-month survivors and 1-month non-survivors.There was no intervention other than normal treatment
  Interventions: Other: This was a retrospective study with no intervention other than normal treatment

INTERVENTIONS:
Other: This was a retrospective study with no intervention other than normal treatment — This was a retrospective study with no intervention other than normal treatment

SUMMARY:
Type A acute aortic dissection (TA-AAD) patients are prone to life-threatening complications and death during the acute phase. Currently, little evidence is available with regards to the relationship between eosinophils (EOS) and TA-AAD.

A total of 274 patients with TA-AAD were eligible for inclusion and 54 patients deceased within 1 month following surgery. Multivariate regression analysis, the general linear model repeated-measures ANOVA analysis (corrected by Greenhouse-Geisser test), receiver-operating characteristics (ROC) curves and a Kaplan-Meier curve were applied for statistical analysis.

DETAILED DESCRIPTION:
For this study, 274 patients with TA-AAD admitted into our hospital between February 2019 and July 2021 were enrolled retrospectively. A total of 54 patients deceased unfortunately within 1 month following surgery. We compared baseline sociodemographic, clinical, and functional status based on the main outcome using t tests or Mann-Whitney U test for continuous data and χ2 or Fisher's exact tests for categorical data. Continuous variables were expressed as mean SD median depending on the normality of distribution, and categorical variables were expressed as absolute number along with their percentages and compared using the chi-square test. Multivariate regression analysis was applied to assess the association between EOS and 1-month mortality in an unadjusted model, in an age-, sex-, Body mass index (BMI)-adjusted model (model 2), adjusted for age, sex, BMI, systolic blood pressure (SBP), diastolic blood pressure (DBP) and mean arterial pressure (MAP) (model 3), and further adjusting for age, sex, BMI, SBP, DBP, MAP, heart rate (HR), diabetes, stroke and hyperlipidemia (model 4). In addition, the general linear model repeated-measures ANOVA analysis (Corrected by Greenhouse-Geisser test in nonspherical cases) was used to compare preoperative EOS and postoperative eight-days EOS. For prognostic analysis, receiver-operating characteristics (ROC) curves were used to determine the optimal cutoff of EOS at different points and the time of postoperative EOS to return to normal levels for the prognostic events. A Kaplan-Meier curve was then applied to compare the prognosis between the 2 subgroups based on the predictive threshold. A P value<0.05 was regarded as statistically significant for all statistical tests.

ELIGIBILITY:
Inclusion Criteria:

* The patients with a diagnosis of Type A acute aortic dissection by the computer tomography

Exclusion Criteria:

* History of cardiogenic shock or cardiac tamponade;
* Iatrogenic aortic dissection;
* Traumatic aortic dissection;
* Severe valvular disease;
* Congenital heart disease;
* Severe organ dysfunction, such as liver and kidney failure;
* Metabolic diseases such as gout or hyperthyroidism;
* Malignant tumor;
* Severe gastrointestinal diseases;
* Recent drug usage that might affect EOS;
* Allergic diseases;
* Infectious diseases;
* Skin diseases;
* Hematological diseases, such as leukemia and myelodysplastic syndromes;
* Immune system diseases.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients were dignosed with Type A acute aortic dissection by the computer tomography between February 2019 and July 2021. A total of 54 patients deceased unfortunately within 1 month following surgery. Depending on mortality within 1 month, the baseline characteristics was compared. Patients were 51.58±11.57 years of age, 203(74.1%) men, and 161(58.8%) with hypertension. There was no discernible difference in gender, BMI, smoking, and alcohol consumption (P>0.05). Moreover, in addition to renal insufficiency, medical histories showed no remarkable deviations between the aforementioned two groups. Non-survivors within 1 month were more likely to have renal insufficiency (6.8% vs. 20.4%; P=0.005).
Sampling Method: Non-Probability Sample
Enrollment: 274 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-04-06 (Actual); Study Completion 2021-06-07 (Actual)

PRIMARY OUTCOMES:
mortality | The first month after operation
  The primary outcome was 1-month mortality

SECONDARY OUTCOMES:
Infection and in-hospital poor prognosis | An average of 1 year
  Poor prognosis was defined as development of any adverse event including organ injury, delirium, cerebral infarction, cerebral hemorrhage and other cardiovascular and cerebrovascular complications.

CONTACTS AND LOCATIONS:
Overall Officials: Yang Yan, Doctor, Study Chair — First Affiliated Hospital Xi'an Jiaotong University
Locations (2):
- China (2):
  - First Affiliated Hospital of Xian JiaotongUniversity, Xi'an, Shaanxi
  - First Affiliated Hospital of Xiann JiaotongUniversity, Xi'an, Shaanxi

REFERENCES:
- [Derived] Wang X, Zhu Y, Ma X, Ren J, Yan Y, Liu Y, Gao H, Zhang S, Chen Y, Yang Y, Deng C. Eosinophil Recovery Time Is Associated with Clinical Outcomes in Patients with Type A Acute Aortic Dissection: a Retrospective Cohort Study. J Cardiovasc Transl Res. 2024 Jun;17(3):723-731. doi: 10.1007/s12265-023-10468-5. Epub 2024 Apr 15. PMID 38622370